CLINICAL TRIAL: NCT00375869
Title: A Prospective Randomized Placebo Controlled Study of the Efficacy and Safety of Darbepoetin Alfa Treatment in Patients With Severe Traumatic Brain Injury
Brief Title: Safety of Darbepoetin Alfa Treatment in Patients With Severe Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Alexandra Hospital (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Demetrios J. Kutsogiannis, MD, MHS, FRCPC, Royal Alexandra Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TBI2006
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Traumatic Brain Injury
Keywords: Neuroprotection; neuron specific enolase; CSF glutamate levels; Darbepoetin Alfa
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Darbepoetin alfa; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darbopoeitin (Active Comparator): The treatment group, comprised of ten patients, will receive an intravenous dose of 200 mcg (1 ml) of darbepoetin (Aranesp®). Patients will be randomly assigned to either the treatment group, or the control group in a 2:1 ratio. The treatment group will be given 200 mcg of darbepoetin intravenously. The control group will be given a matching placebo of 1 mL of normal saline.
  Interventions: Drug: Darbeopoetin
- Normal Saline (Placebo) (Placebo Comparator): The treatment group, comprised of ten patients, will receive an intravenous dose of 200 mcg (1 ml) of darbepoetin (Aranesp®). Patients will be randomly assigned to either the treatment group, or the control group in a 2:1 ratio. The treatment group will be given 200 mcg of darbepoetin intravenously. The control group will be given a matching placebo of 1 mL of normal saline.
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Darbeopoetin — The treatment group, comprised of ten patients, will receive an intravenous dose of 200 mcg (1 ml) of darbepoetin (Aranesp®). Patients will be randomly assigned to either the treatment group, or the control group in a 2:1 ratio. The treatment group will be given 200 mcg of darbepoetin intravenously. The control group will be given a matching placebo of 1 mL of normal saline.
  Other Names: ARANESP
  Arms: Darbopoeitin
Drug: Normal Saline (Placebo) — The treatment group, comprised of ten patients, will receive an intravenous dose of 200 mcg (1 ml) of darbepoetin (Aranesp®). Patients will be randomly assigned to either the treatment group, or the control group in a 2:1 ratio. The treatment group will be given 200 mcg of darbepoetin intravenously. The control group will be given a matching placebo of 1 mL of normal saline.
  Other Names: Placebo
  Arms: Normal Saline (Placebo)

SUMMARY:
The purpose of this study is to see if the treatment of severely brain injured patients with darbepoetin (a long acting form of erythropoietin) will be safe, and will reduce brain damage by decreasing harmful levels of chemicals in the brain.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a common neurosurgical problem with a high morbidity and mortality. Studies interested in defining possible therapeutic targets in TBI have led to an appreciation of two phases of injury. These phases are referred to as primary and secondary TBI. The primary injury encompasses the immediate insult, diffuse axonal injury, hemorrhage, contusion, and primary ischemia. The secondary injury evolves over the post-traumatic period and is due to a combination of vasogenic and cytotoxic edema resulting from several processes including; glutamate excitotoxicity, disturbance of ionic homeostasis, lipid peroxidation, generation of nitric oxide (NO) and free radicals, and release of inflammatory regulators such as bradykinin and eicosanoids. It has long been recognized that one of the most important factors in the secondary injury process is the indiscriminate release of the excitatory neurotransmitter glutamate from neurons and glia. Glutamate excitotoxicity leads to substantial intraneuronal release of calcium which in turn mediates the activation of phospholipases which generate arachadonic acid, the activation of proteases, and the activation of NO, all of which cause neuronal membrane disruption and loss of ionic equilibrium. Receptors for erythropoietin (EPOr) are distributed throughout the brain and studies have demonstrated that these receptors are not only important in the process of development but also in neuroprotection. Treatment with erythropoietin (EPO) protects neurons in models of ischemic and traumatic degenerative damage due to exocitotoxins and consequent generation of free radicals including NO. EPOr activation also prevents the indiscriminate exocytosis of glutamate in a model of chemically induced ischemia on neurons of rat hippocampus.

The hypothesis of this study is that treatment of severely brain injured patients with darbepoetin alfa (Aranesp®) will be safe and reduce the cerebrospinal fluid (CSF) levels of glutamate within a 96 hour period after traumatic brain injury. This effect is potentially mediated through the activation of EPO receptors whose activation prevents the exocytosis of glutamate, a known neurocytotoxin, into CSF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 inclusive.
* Admitted to ICU with a TBI and a GCS ≤ 8 with a motor score < 6.
* Patient must have a functioning external ventricular drain in place for intracranial pressure (ICP) monitoring.
* Completion of informed consent by the next-of-kin or legal guardian.
* Randomization within 12 hours of initial triage by medical or paramedical staff.
* Abnormal CT of the brain.

Exclusion Criteria:

* Pregnancy
* Cardiac arrest during the current hospital admission.
* Bilateral non-reactive dilated pupils at the time of randomization.
* A history of renal failure, NYHA class IV congestive heart failure, or recent myocardial infarction (within 6 months).
* A history of primary or secondary polycythemia.
* Previous adverse reactions to rhEPO or darbepoetin.
* Previous history of seizure disorder.
* Recent history (within the past 3 months) of significant uncontrolled hypertension defined as SBP > 200 mm Hg or DBP > 110 mmHg.
* Patients involved in other clinical investigations involving therapeutic interventions
* Hemoglobin ≥150 g/L in females
* Hemoglobin ≥160g/L in males
* Past history of thrombotic events

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Neuron-specific serum enolase, CSF glutamate and CSF S100B levels in patients receiving darbepoetin compared to placebo | over 96 hours
  The primary outcome measures include Neuron-specific serum enolase, CSF glutamate and CSF S100B levels in patients receiving darbepoetin compared to placebo over a 96 hour period and ICP levels in patients receiving darbepoetin compared to placebo over a 96 hour period

SECONDARY OUTCOMES:
Secondary outcome measures include ICU and hospital length of stay, GCS at ICU discharge, survival status, location after ICU and hospital discharge. GCS will be evaluated at day 28 and 1 year. | day 28 and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Demetrios J. Kutsogiannis, MD MHS FRCPC, Principal Investigator — Division of Critical Care Medicine
Locations (2):
- Canada (2):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta